CLINICAL TRIAL: NCT06252623
Title: A Human Laboratory Study of Exenatide for Reducing the Reinforcing Effects of Cocaine
Brief Title: Exenatide For Reducing the Reinforcing Effects of Cocaine
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was closed due to the inability to acquire the study drug.
Sponsor: Christopher D. Verrico (Other)
Responsible Party: Sponsor-Investigator, Christopher D. Verrico, Associate Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-52307
Record Dates: First submitted 2024-01-29; First posted 2024-02-12 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Cocaine Use Disorder
Keywords: cocaine; GLP-1; exenatide; cocaine use disorder
MeSH Terms: interventions — Exenatide; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Drug: Exenatide 2 mg [Bydureon] (Experimental): Participants will receive once-weekly subcutaneous exenatide (2 mg) injections for 6 weeks.
  Interventions: Drug: Exenatide
- Drug: Placebo (Placebo Comparator): Participants will receive once-weekly subcutaneous saline (i.e., placebo) injections for 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exenatide — Exenatide will be purchased commercially as Bydureon® for subcutaneous injection and administered at 2 mg once a week for 6 weeks. Each single-dose, dual-chamber pen contains 0.65 mg of diluent and 2 mg of exenatide, which remains isolated until mixed.
  Other Names: Bydureon
  Arms: Drug: Exenatide 2 mg [Bydureon]
Drug: Placebo — Sterile saline will be used as the placebo and administered subcutaneously once a week for 6 weeks.
  Other Names: saline
  Arms: Drug: Placebo

SUMMARY:
This study will determine the safety and tolerability of exenatide (Bydureon®) as a pharmacotherapy for cocaine use disorder. An inpatient human laboratory study will be conducted in which the self-administration of cocaine, as well as the subjective and physiological effects of cocaine, are evaluated during maintenance on placebo and exenatide.

Although exenatide (Bydureon) is approved by the Food and Drug Administration (FDA) for the treatment of type 2 diabetes, it has not been approved by the FDA to treat cocaine use; therefore, it is called an investigational drug.

DETAILED DESCRIPTION:
Cocaine (COC) use disorder (CUD) remains a significant medical, social, and legal concern. According to the 2019 National Survey on Drug Use and Health, approximately 1 million Americans meet the criteria for CUD. Behavioral therapies, such as cognitive-behavioral therapy (CBT), are the mainstay of current treatment approaches for CUD. However, because CBT alone has limited efficacy, the identification and development of pharmacotherapy that enhances the effectiveness of CBT is a high priority. Therefore, developing evidence-based interventions to reduce adverse outcomes associated with drug use and support the long-term recovery of people following treatment are top priorities for National Institute on Drug Abuse (NIDA) research. To that end, NIDA supports a dual strategy to accelerate medication development for CUD: (1) translating preclinical knowledge to target novel pathways and circuits and (2) repurposing medications already approved for other indications.

There is now substantial preclinical evidence that glucagon-like peptide-1 (GLP-1) receptor (GLP-1R) agonists attenuate behaviors that model both the consumption and seeking of highly palatable food and several commonly abused drugs, including alcohol, cocaine, and nicotine. The neurobiological mechanisms underlying food intake and drug-seeking overlap to a degree. Homeostatic and hedonic pathways regulate food intake. The homeostatic pathway regulates energy balance, while the hedonic pathway can override homeostatic regulation during periods of relative energy abundance, increasing the desire to consume highly palatable foods. In the homeostatic pathway, food intake stimulates the production and secretion of incretin hormones and satiation factors, like GLP-1, via both intestinal L-cells and neurons in the nucleus of the solitary tract (NTS). GLP-1-producing neurons of the NTS project to the arcuate nucleus (ARC) of the hypothalamus. In the ARC, GLP-1R activation suppresses feeding by activating anorexigenic neurons, which contain cocaine- and amphetamine-regulated transcript (CART), and inhibiting orexigenic neurons. NTS neurons also project to the ventral tegmental area (VTA), the nucleus accumbens (NAc), the laterodorsal tegmental nucleus (LDT), and the lateral septum. GLP-1 binding, messenger ribonucleic acid (mRNA), and immunoreactivity are detected in these same areas, as well as on VTA projections to the NAc and LDT projections to both the NAc and VTA. Direct activation of GLP-1R in the VTA,[10] NAc, LDT, or the lateral septum decreases palatable food intake, underscoring the critical role of GLP-1 in regulating the hedonic value of food.

The overall objective of this application is to determine if GLP-1R agonism is a viable treatment strategy for CUD. This goal will be achieved through the conduct of a rigorous human clinical pharmacology study in which non-treatment-seeking COC users (n=44) will be randomized (1:1) to placebo or extended-release (XR) exenatide (i.e., exenatide dose is a between-subject factor) for six weeks. The 6-week maintenance period, sufficient to achieve steady-state, will result in more stable concentrations of clinically effective doses before assessing treatment effects. Before and after the 6-week maintenance period, the investigators will determine COC (0, 20, 40 mg: IV) self-administration rates. To accurately predict clinical efficacy, the investigators will use forced-choice procedures in which participants choose to either self-administer COC or receive money.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking
2. Male or female ≥ 18 and ≤ 65 years of age
3. Willing and able to provide written informed consent and participate in all required study activities
4. Self-reported recent use of smoked or IV COC verified by a COC positive urine (≥ 150 ng/mL)
5. Report using COC for ≥ 10 years and using ≥ 2 grams of COC/week
6. Have vital signs as follows, resting pulse between 50 and 95 bpm, blood pressure (BP) between 90-150 mmHg systolic and 45-95 mmHg diastolic.
7. Have hematology and chemistry laboratory tests that are within reference limits (±10%), with the following exception, pancreatic tests (lipase and amylase) must be within normal limits
8. Have a medical history, physical examination, electrocardiogram (ECG), drug-use history, and the Mini-International Neuropsychiatric Interview (M.I.N.I.) demonstrating no clinically significant contraindications for study participation, in the judgment of a Study Physician and the Principal Investigator.
9. Agree (if the subject is female and of child-bearing potential) to use at least one of the following methods of birth control from time of the first administration of the study drug to at least 7 days post the last dose of study drug, unless the partner is surgically sterile (underwent vasectomy),

   1. oral contraceptives,
   2. contraceptive sponge,
   3. patch,
   4. double barrier (diaphragm/spermicidal or condom/spermicidal),
   5. intrauterine contraceptive system,
   6. etonogestrel implant,
   7. medroxyprogesterone acetate contraceptive injection,
   8. complete abstinence from sexual intercourse, and/or
   9. hormonal vaginal contraceptive ring
10. Women of child-bearing potential must provide negative urine pregnancy tests prior to randomization, and at study visits as indicated in the Research Strategy
11. No contraindications/allergies to COC or exenatide
12. Cardiovascular and subjective responses to COC within acceptable

Exclusion Criteria:

1. Clinically significant medical conditions .
2. Meet diagnostic criteria for substance-use disorders other than for CUD that in the opinion of the study physician would comprise the well-being of the participant.
3. Seeking treatment for a substance use disorder.
4. Any laboratory test deemed clinically significant by the study physician.
5. Type 1 or type 2 Diabetes Mellitus (HbA1C level of ≥6.5%)
6. Previous medically adverse reaction to the study medications (Bydureon) or COC.
7. Medication use that might interact with COC or exenatide, or otherwise compromise safety.
8. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2.
9. Severe cardiovascular disease (history of myocardial infarction, life-threatening arrhythmia, or worsening angina pectoris).
10. Severe gastrointestinal disease (i.e., severe gastroparesis).
11. Previous history of pancreatitis or risk of pancreatitis.
12. Creatinine clearance <45 or end stage renal disease (ESRD).
13. Contraindications to treatment with exenatide (e.g., personal of family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type-2; history of pancreatitis or risk of pancreatitis).
14. Participation in a clinical trial within 30 days of admission.
15. Positive urine pregnancy test or females trying to conceive, donated ova, are pregnant, or are lactating or breast feeding at screening or throughout study.
16. Positive urine screen for drugs-of-abuse, other than COC or marijuana, or breath alcohol test. Note, if positive for opioids or oxycodone but recent opioid use for acute pain is reported by the subject, then the subject can be included at the discretion of the Primary Investigator and/or Study Physician.
17. Have a history of suicidal ideation.
18. Have any illness or condition which in the opinion of the Principal Investigator and/or the Study Physician would preclude safe and/or successful completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of up to 10 active cocaine doses | 6 weeks
  The primary outcome measure will be the proportion of up to 10 active cocaine doses (i.e., 20 and 40 mg) self-administered post-treatment.
Subjective Effects | 6 weeks
  Subjective effects produced by cocaine or placebo will be measured using a visual analog scale (VAS) form. Visual analog scales rely on a visual cue (a ten-centimeter horizontal line anchored with the phrases "0 - not at all" to "100 - extremely") to evaluate the subjective effects of amphetamine. Instructions require that patients bisect the line at the point matching their "current" subjective states after ingesting a substance.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | 6 weeks
  Safety will be assessed by recording severity and number of treatment-emergent adverse events (TEAEs), which will be analyzed over the entire treatment and follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Verrico, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No